CLINICAL TRIAL: NCT03618823
Title: Randomized Clinical Trial of Non-Opioid Pain Medications After Adenotonsillectomy
Brief Title: Non-opioids for Analgesia After Adenotonsillectomy in Children
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Early termination due to COVID-19 cases and cancelled surgeries.
Sponsor: David Chi, MD (Other)
Responsible Party: Sponsor-Investigator, David Chi, MD, Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19040036 (Part 1)
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2021-11-10 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-10

CONDITIONS: Adenotonsillectomy; Post-operative Analgesia; Opioid Use
Keywords: analgesia; pain control; adenotonsillectomy; tonsillectomy; opioids; post-operative pain
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Oxycodone; Ibuprofen; Acetaminophen

STUDY DESIGN:
Intervention Model Description: Experimental, open-label randomized control trial.
Masking Description: Open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Opioid pain control (Experimental): Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary.
  Interventions: Drug: Oxycodone; Drug: Ibuprofen; Drug: Acetaminophen
- Non-opioid pain control (Active Comparator): Patients in this group will be receiving therapy for pain control with acetaminophen and ibuprofen only. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the diary.
  Interventions: Drug: Ibuprofen; Drug: Acetaminophen

INTERVENTIONS:
Drug: Oxycodone — Oxycodone will be prescribed at a dose in the range of 0.025 mg/kg to 0.10 mg/kg every four hours or as needed for adequate pain management. The total supply will be limited to seven days. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
  Arms: Opioid pain control
Drug: Ibuprofen — Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.
Drug: Acetaminophen — Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours. It will be prescribed in liquid suspension form for ease of use in pediatric populations. Subjects or parents will purchase this medication and dosage will be given to subjects in easy-to-understand language.

SUMMARY:
The goal of this study is to determine if non-opioid pain control is a safe way to manage pain after adenotonsillectomy surgery in children. The investigators will be randomly assigning children aged 3-17 to one of two groups: one group will receive non-opioid pain medication only, and the other group will receive opioid and non-opioid medications for pain control. The investigators will analyze the data and determine if there is a difference in pain control between the two drug regimens, and if there are any other associated complications between the two groups.

This study is important because if we can demonstrate that there is little difference in outcomes and pain control between the two groups, a strong argument can be made for reducing or eliminating opioid prescription after adenotonsillectomy. This may protect future children from the risks of taking opioid medications and help to reduce the scope of the opioid epidemic.

DETAILED DESCRIPTION:
Purpose: To determine if non-opioid pain control is a safe and effective option in the treatment of post-operative pain following adenotonsillectomy in various pediatric age groups.

Methods: The subject population will be patients between the ages of 3 and 17 who will undergo adenotonsillectomy. The study will consist of two unblinded arms - patients receiving standard pain control regimen which include opioids and non-opioids, and patients receiving non-opioid pain medications only. In the diary they will receive, patients or caregivers will record quantity and dosage of pain medication taken each day, a survey, and pain ratings measured by the Wong-Baker FACES Pain Rating Scale. Within 4-8 weeks post-operatively the patients will return for a follow up appointment along with their diary. Demographic information such as age, race, gender, household income will be extracted from the diary and the electronic medical record. Information such as surgical technique, concurrent operations, post-operative pain prescription (types, weight based dosage, and total days prescribed) will be extracted from the electronic medical record and recorded as well. Outcomes measured will include pain scale rating and rates of complications between the two groups.

Significance: If it can be demonstrated that non-opioid pain control after adenotonsillectomy does not lead to increased pain or worse outcomes in certain pediatric age groups, a strong argument can be made for the cessation of opioid prescription for these ages following adenotonsillectomy. Given the widespread opioid epidemic, this would be a significant step in curbing the massive opioid problem, as well as reducing the adverse effects of opioid usage in pediatric populations.

ELIGIBILITY:
Inclusion Criteria:

• Patients age 3 - 17 undergoing adenotonsillectomy

Exclusion Criteria:

* Down syndrome
* History of coagulopathy
* Craniofacial abnormalities
* Caregivers who cannot speak, read, or write in English proficiently
* Patients who take opioids during the enrollment period
* Patients who take chronic opioids
* Pregnancy
* Allergy to or contraindication for taking any of the study medications
* Patients who have the inability to communicate
* Patients who have the inability to localize pain

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 268 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-05-18 (Actual); Study Completion 2020-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David H Chi, MD, Principal Investigator — Clinical Director, Division of Pediatric Otolaryngology, Children's Hospital of Pittsburgh
Locations (1):
- UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Only co-investigators as listed under the University of Pittsburgh IRB (Institutional Review Board) protocol for this study will have access to all data and analysis. Data will be shared via UPMC-associated OneDrive and will only be shared between these investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be maintained for at least 7 years or until the child turns 23 per University of Pittsburgh policy.
Access Criteria: All data will be shared as-needed for analysis amongst the listed co-investigators in the University of Pittsburgh IRB protocol for this study. It will be stored on the UPMC OneDrive.

REFERENCES:
- [Background] Van Cleve WC, Grigg EB. Variability in opioid prescribing for children undergoing ambulatory surgery in the United States. J Clin Anesth. 2017 Sep;41:16-20. doi: 10.1016/j.jclinane.2017.05.014. Epub 2017 Jun 3. PMID 28802595
- [Background] Rudd RA, Seth P, David F, Scholl L. Increases in Drug and Opioid-Involved Overdose Deaths - United States, 2010-2015. MMWR Morb Mortal Wkly Rep. 2016 Dec 30;65(50-51):1445-1452. doi: 10.15585/mmwr.mm655051e1. PMID 28033313
- [Background] Schuchat A, Houry D, Guy GP Jr. New Data on Opioid Use and Prescribing in the United States. JAMA. 2017 Aug 1;318(5):425-426. doi: 10.1001/jama.2017.8913. No abstract available. PMID 28687823
- [Background] Feinberg AE, Chesney TR, Srikandarajah S, Acuna SA, McLeod RS; Best Practice in Surgery Group. Opioid Use After Discharge in Postoperative Patients: A Systematic Review. Ann Surg. 2018 Jun;267(6):1056-1062. doi: 10.1097/SLA.0000000000002591. PMID 29215370
- [Background] Monitto CL, Hsu A, Gao S, Vozzo PT, Park PS, Roter D, Yenokyan G, White ED, Kattail D, Edgeworth AE, Vasquenza KJ, Atwater SE, Shay JE, George JA, Vickers BA, Kost-Byerly S, Lee BH, Yaster M. Opioid Prescribing for the Treatment of Acute Pain in Children on Hospital Discharge. Anesth Analg. 2017 Dec;125(6):2113-2122. doi: 10.1213/ANE.0000000000002586. PMID 29189368
- [Background] Holte K, Kehlet H. Effect of postoperative epidural analgesia on surgical outcome. Minerva Anestesiol. 2002 Apr;68(4):157-61. PMID 12024074
- [Background] van Boekel RLM, Warle MC, Nielen RGC, Vissers KCP, van der Sande R, Bronkhorst EM, Lerou JGC, Steegers MAH. Relationship Between Postoperative Pain and Overall 30-Day Complications in a Broad Surgical Population: An Observational Study. Ann Surg. 2019 May;269(5):856-865. doi: 10.1097/SLA.0000000000002583. PMID 29135493
- [Background] Bean-Lijewski JD, Kruitbosch SH, Hutchinson L, Browne B. Post-tonsillectomy pain management in children: can we do better? Otolaryngol Head Neck Surg. 2007 Oct;137(4):545-51. doi: 10.1016/j.otohns.2007.06.731. PMID 17903568
- [Background] Luk LJ, Mosen D, MacArthur CJ, Grosz AH. Implementation of a Pediatric Posttonsillectomy Pain Protocol in a Large Group Practice. Otolaryngol Head Neck Surg. 2016 Apr;154(4):720-4. doi: 10.1177/0194599815627810. Epub 2016 Feb 16. PMID 26884362
- [Background] Kelly LE, Sommer DD, Ramakrishna J, Hoffbauer S, Arbab-Tafti S, Reid D, Maclean J, Koren G. Morphine or Ibuprofen for post-tonsillectomy analgesia: a randomized trial. Pediatrics. 2015 Feb;135(2):307-13. doi: 10.1542/peds.2014-1906. PMID 25624387
- [Derived] Whelan RL, McCoy JL, Mirson L, Maguire RC, Jabbour N, Simons JP, Dohar JE, Kitsko DJ, Stapleton AL, Tobey ABJ, Alper CM, Shaffer AD, Bennett ZR, Chi DH. Opioid Analgesia Following Pediatric Adenotonsillectomy: A Randomized Clinical Trial. Otolaryngol Head Neck Surg. 2025 Aug;173(2):392-401. doi: 10.1002/ohn.1280. Epub 2025 May 21. PMID 40396501

RESULTS

PARTICIPANT FLOW:
Groups:
- Opioid Pain Control: Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary.
  Oxycodone: Oxycodone will be prescribed at a dose in the range of 0.025 mg/kg to 0.10 mg/kg every four hours or as needed for adequate pain management. The total supply will be limited to seven days. It will be prescribed in liquid suspension form for ease of use in pediatric populations.
  Ibuprofen: Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses.
  Acetaminophen: Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours.
- Non-opioid Pain Control: Patients in this group will be receiving therapy for pain control with acetaminophen and ibuprofen only. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the diary.
  Ibuprofen: Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses.
  Acetaminophen: Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours.
Period: Overall Study
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Started | 132 | 136
Completed | 69 | 75
Not Completed | 63 | 61
Not completed — Lost to Follow-up | 63 | 61

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid Pain Control | Non-opioid Pain Control | Total
Number analyzed (Participants) | 132 | 136 | 268
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.39 (3.33) | 8.15 (3.33) | 8.27 (3.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 | 68 | 137
  Male | 63 | 68 | 131
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 5 | 6
  Not Hispanic or Latino | 127 | 120 | 247
  Unknown or Not Reported | 4 | 11 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 9 | 11 | 20
  White | 118 | 120 | 238
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 2 | 3 | 5
BMI Centile [Mean (Standard Deviation); unit: Percentage] | 66.42 (32.81) | 67.20 (31.44) | 66.81 (32.06)

OUTCOME MEASURES:

1. Primary Outcome: Average Pain Burden
Description: Average pain over 14 post-operative days before and after medications. This is quantified using the validated Wong-Baker FACES pain metric. Patients receive a take-home pain diary and for 14 days report their maximum pain both before and after taking pain medication. The mean of these pain ratings will be the primary outcome measure. The Wong-Baker FACES scale is from 0 (min) to 10 (max). A higher score indicates worse outcome/pain.
Time Frame: 14 days post-operatively
Population: Participants were analyzed for average pain burden if they completed the take-home pain diary and pain scores were recorded.
Measure: Mean (Standard Error); unit: Score on a scale
Groups:
- Opioid Pain Control Group: Patients in this group will be receiving triple therapy for pain control with oxycodone, acetaminophen, and ibuprofen. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the pain diary.
  Oxycodone: Oxycodone will be prescribed at a dose in the range of 0.025 mg/kg to 0.10 mg/kg every four hours or as needed for adequate pain management. The total supply will be limited to seven days. It will be prescribed in liquid suspension form for ease of use in pediatric populations.
  Ibuprofen: Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses.
  Acetaminophen: Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours.
- Non-opioid Pain Control Group: Patients in this group will be receiving therapy for pain control with acetaminophen and ibuprofen only. They will be asked to complete a pain diary which will be used to determine the level of pain control achieved with this regimen. The diary will be completed by post-operative day 14. A post-operative appointment between 4-8 weeks will be scheduled and the patient and caregiver will return the diary.
  Ibuprofen: Ibuprofen will be prescribed at 10 mg/kg to be taken every 6 hours for the first three post-operative days. After the first three days, the subject should take the ibuprofen every 6 hours as needed for pain control. The daily dose of ibuprofen is not to exceed 1200mg or more than 4 individual doses.
  Acetaminophen: Acetaminophen will be prescribed at 15mg/kg to be taken every 4 hours for the first three days, except when sleeping. After the first three days, the subject should take the acetaminophen every 4 hours as needed for pain control. The daily dose of acetaminophen is not to exceed 5 doses in 24 hours.
Arm/Group | Opioid Pain Control Group | Non-opioid Pain Control Group
Number analyzed (Participants) | 60 | 68
Score on a scale
  Before | 5.78 (0.25) | 5.66 (0.23)
  After | 2.33 (0.22) | 2.24 (0.21)
Statistical Analysis 1: Comparison: Opioid Pain Control Group vs Non-opioid Pain Control Group; There will be no difference in pain scores between opioid and non-opioid groups from before medication to after while controlling for total duration of mediation use (duration mean=10.11 days); Test type: Equivalence — All pain scores were included due to the sample size. Alpha =.05 Power = .80 Desired effect size of 0.30 Size of n=145 in each group was determined, however this was not reached for sufficient power; p = .912, Mixed Models Analysis; Two-way mixed-model analysis of variance

2. Secondary Outcome: Number of Participants With ED (Emergency Department) or Urgent Care Visits
Description: Number of participants with emergency department or urgent care visits in 14 post-operative days - assessed via the electronic medical record and the take-home pain diary.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants | 8 | 11
Statistical Analysis 1: Comparison: Opioid Pain Control vs Non-opioid Pain Control; There will be no difference in ED (Emergency Department) or urgent care visits between opioid and non-opioid pain control groups; Test type: Superiority; p = .630, Fisher Exact; Odds Ratio (OR) = 1.311, 95% CI 2-sided [.494 to 3.478]

3. Secondary Outcome: Number of Side Effects of Medications
Description: Number of any of the following side effects experienced: Nausea, vomiting, constipation, stomach ache, difficulty breathing. Assessed at follow-up and take-home pain diary.
Time Frame: 14 days post-operatively
Population: Participants were analyzed for side effects of medications if they completed the take-home pain diary and side effects of medications were recorded.
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 65 | 66
Participants
  0 side effect | 38 | 35
  1 side effect | 10 | 22
  2 side effect | 7 | 7
  3 side effect | 9 | 2
  4 side effect | 1 | 0
  5 side effect | 0 | 0

4. Other Pre Specified Outcome: Number of Participants With Readmissions
Description: Number of participants with hospitalizations after discharge in 14 days - assessed using the electronic medical record and the take-home pain diary.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants | 3 | 8

5. Other Pre Specified Outcome: Average Dose of Each Analgesic Used
Description: In the take-home pain diary, patients will record the amount of medication taken for each dose. The mean value of these doses will be calculated and averaged within each group to determine the average dose of each analgesic used.
Time Frame: 14 days post-operatively
Population: Participants who took mg dose instead of ml for acetaminophen and ibuprofen were taken out of the analysis.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 61 | 67
Milliliters
  Acetaminophen | 6.54 (2.87) | 7.52 (6.47)
  Ibuprofen | 7.53 (4.08) | 7.53 (4.74)
  Oxycodone | 0.13 (0.19) | 0.04 (0.24)

6. Other Pre Specified Outcome: Duration of Each Analgesic Used
Description: Using the results of the take-home pain diary, we will calculate the average number of days of use of each analgesic for each group. The last day after which there is no subsequent use of analgesic will define the end-point of the duration of use.
Time Frame: 14 days post-operatively
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
days
  Acetaminophen | 8.61 (2.97) | 8.64 (3.40)
  Ibuprofen | 8.49 (3.42) | 8.75 (3.46)
  Oxycodone | 2.62 (2.90) | 0.45 (1.66)

7. Other Pre Specified Outcome: Mean of Total Quantity of Pain Medications Taken
Description: Using the take-home pain diary, the total amount in mL of each analgesic used over 14 days by each patient in a group will be averaged and reported.
Time Frame: 14 days post-operatively
Population: Participants who took mg dose instead of ml for acetaminophen and ibuprofen were taken out of the analysis.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 61 | 67
Milliliters
  Acetaminophen | 292.48 (178.73) | 326.98 (269.66)
  Ibuprofen | 324.14 (225.70) | 334.65 (234.18)
  Oxycodone | 6.47 (9.89) | 2.96 (14.84)

8. Other Pre Specified Outcome: Overall Pain Relief Satisfaction
Description: Score assigned by the patient at the end of 14 post-operative days in the take-home pain diary using a Likert scale. Patients will respond to the following statement "I am happy with the pain relief I received in the last 14 days" with responses ranging from strongly agree to strongly disagree. The responses will be assigned a numerical value, from 0 (strongly disagree) to 4 (strongly agree), and the average value for all subjects in the group will be reported as the overall pain relief satisfaction. Higher scores mean a better outcome.
Time Frame: 14 days post-operatively
Population: Participants were analyzed for overall pain relief satisfaction if they completed the take-home pain diary and overall pain relief satisfaction was recorded.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 63 | 64
score on a scale | 3.35 (0.79) | 3.09 (0.96)

9. Other Pre Specified Outcome: Post-operative Nursing Phone Calls
Description: Number of post-operative phone calls to nursing staff, obtained using the electronic medical record.
Time Frame: 14 days post-operatively
Measure: Mean (Standard Deviation); unit: post-operative phone calls
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
post-operative phone calls | 0.35 (0.66) | 0.47 (0.79)

10. Other Pre Specified Outcome: Number of Night-time Awakenings
Description: Number of night-time awakenings reported in 14 days - assessed via the take-home pain diary.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants
  None | 10 | 13
  Some nights (1-4) | 33 | 28
  Many nights (5-9) | 19 | 18
  Most nights (10-14) | 3 | 7
  No response | 4 | 9

11. Other Pre Specified Outcome: Non-opioid Group Switching to Opioid Group
Description: Number of non-opioid group members switching to receiving opioid medication - assessed via the take-home pain diary.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Non-opioid Pain Control
Number analyzed (Participants) | 75
Participants | 7

12. Other Pre Specified Outcome: Need for Follow-up Appointment
Description: Does the parent/guardian believe his/her child would require a follow-up appointment - assessed using the individual pain diary.
Time Frame: two months post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants
  No response | 7 | 11
  No | 54 | 49
  Yes | 8 | 15

13. Other Pre Specified Outcome: Household Income
Description: Total household income ranges will be assessed in the take-home pain diary and reported.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants
  No response | 14 | 13
  $0-25,000 | 2 | 7
  $25,001-50,000 | 8 | 7
  $50,001-75,000 | 9 | 11
  $75,001-100,000 | 11 | 9
  $100,001-125,000 | 9 | 6
  $125,001-150,000 | 3 | 3
  $150,001-175,000 | 1 | 1
  $175,001-200,000 | 7 | 5
  $200,000 or more | 2 | 2
  Prefer not to answer | 3 | 11

14. Other Pre Specified Outcome: Education Level
Description: Using the take-home pain diary, parents/guardians of the patients will identify the highest level of education achieved by anyone in the household.
Time Frame: 14 days post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
Number analyzed (Participants) | 69 | 75
Participants
  No response | 14 | 13
  Some high school | 0 | 3
  High school degree | 4 | 8
  Vocational or associate degree | 7 | 10
  Some college | 7 | 4
  College degree | 18 | 24
  Master's degree | 14 | 9
  Professional or academic doctorate | 4 | 3
  Prefer not to answer | 1 | 1

ADVERSE EVENTS:
Time Frame: 5-9 weeks depending on the date of the follow-up appointment
Description: Number of participants at risk for adverse events was based on treatment received. The number started in the participant flow was based on group assignment.
  17 of the 136 participants who were assigned to the non-opioid group received an opioid prescription upon parental request.
  The number of participants at risk in the opioid group were 149 (132 assigned + 17 cross-over to opioid).
  The number of participants at risk in the non-opioid group were 119 (136 assigned - 17 cross-over).
Arm/Group | Opioid Pain Control | Non-opioid Pain Control
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/119
Serious Adverse Events (participants affected / at risk) | 9/149 | 4/119
Other Adverse Events (participants affected / at risk) | 38/149 | 22/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid Pain Control (N=149) | Non-opioid Pain Control (N=119)
Post-Tonsillectomy Hemorrhage Requiring Operative Intervention (Surgical and medical procedures) | 7 | 3
Dehydration Requiring Inpatient Admission (General disorders) | 2 | 0
Oxygen Desaturation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Oxygen desaturation requiring prolongation of hospitalization for tonsillectomy and adenoidectomy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Opioid Pain Control (N=149) | Non-opioid Pain Control (N=119)
Post-Tonsillectomy Hemorrhage Not Requiring Operative Intervention (Vascular disorders) | 13 | 8
Emergency Department Visit for Pain (General disorders) | 8 | 0
Nursing Phone Call for Pain (General disorders) | 23 | 15
Nausea or Vomiting (General disorders) | 10 | 3

LIMITATIONS AND CAVEATS:
Early termination due to COVID-19 cases and cancelled surgeries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-19): https://cdn.clinicaltrials.gov/large-docs/23/NCT03618823/Prot_SAP_000.pdf